CLINICAL TRIAL: NCT02774837
Title: Open Label Study of Nucleus(t)Ide Treated Patients Randomised to Tenofovir, or Tenofovir + Telbivudine
Brief Title: Tenofovir Versus Tenofovir + Telbivudine for Chronic Hepatitis B
Acronym: DUAL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seng Gee Lim (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government); Singapore Clinical Research Institute (Other)
Responsible Party: Sponsor-Investigator, Seng Gee Lim, Director of Hepatology, National University Health System, Singapore
Organization: National University Health System, Singapore (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/00215
Record Dates: First submitted 2016-05-12; First posted 2016-05-17 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Chronic Hepatitis B
Keywords: nucleoside analogues; tenofovir; telbivudine; quantitative HBsAg; combination therapy
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir; Telbivudine

STUDY DESIGN:
Intervention Model Description: Two arm parallel study
Oversight: Data Monitoring Committee: No

ARMS (2):
- combination (Experimental): Tenofovir disoproxil oral tablets 300mg once daily for 96 weeks and Telbivudine 600mg oral tablets once daily for 96 weeks
  Interventions: Drug: Tenofovir disoproxil; Drug: Telbivudine
- mono therapy (Active Comparator): Tenofovir disoproxil oral tablets 300mg once daily for 96 weeks
  Interventions: Drug: Tenofovir disoproxil

INTERVENTIONS:
Drug: Tenofovir disoproxil — Tenofovir disoproxil 300mg once daily for 96 weeks
  Other Names: Viread
Drug: Telbivudine — Telbivudine oral tablets 600mg once daily for 96 weeks
  Other Names: Sebivo
  Arms: combination

SUMMARY:
Chronic Hepatitis B is the most common cause of chronic viral liver disease worldwide afflicting 350 million persons, leading to significant morbidity and mortality due to liver disease and HCC in 20-40% of infected persons. With the advent of nucleoside analogues, this rescued patients with significant risk of disease progression, but in most circumstances, therapy was needed long term as HBsAg seroclearance was an uncommon occurrence, and stopping therapy was associated with relapse of disease and hepatitis B flares. The use of pegylated interferons showed increased HBeAg seroconversion and HBsAg seroclearance rates compared to nucleoside analogues , however combination nucleos(t)ide analogue therapy has been quite disappointing. However a recent showed that the combination of telbivudine and tenofovir in a response guided therapy design, had a remarkable 6% HBsAg seroclearance at week 52 in patients. Such results require further confirmation. There is currently an unmet need for the large number of patients on long term nucleoside analogue therapy who have not achieved HBeAg seroconversion or HBsAg seroclearance. Such patients are seeking alternatives to long term therapy hence an exploration of other therapeutic strategies is attractive. An additional benefit of telbivudine has been the surprising improvement in renal function and this study seeks to examine whether this can improve the renal impairment that may be seen with tenofovir. Our study proposes to examine if the combination of tenofovir and telbivudine can improve endpoints. Patients fulfilling inclusion and exclusion criteria will be randomized to tenofovir or tenofovir and telbivudine (1:1 ratio). The primary endpoint will be a qHBsAg reduction of >1log at week 96, which may predict future HBsAg seroclearance, which is also a secondary endpoint. An additional primary endpoint is increase in eGFR in the combination arm compared to the monotherapy arm. The study aims to enroll 146 patients randomized 1:1 ratio (73:73) patients. Multivariate analysis will be performed of baseline and on-treatment factors that predict the primary outcome.

DETAILED DESCRIPTION:
Each subject must sign and date a study-specific informed consent form (ICF) prior to their participation in any screening activities. Prospective subjects should be screened no more than 28 days prior to administration of the first dose of study drug on Day 1. Screening evaluations will be used to determine eligibility of each candidate for study enrollment. Subjects meeting all of the inclusion criteria and none of the exclusion criteria as determined during screening will be eligible for the study. Candidates who fail to meet eligibility criteria by screening evaluations may be re-screened one time. Eligible patients at the end of screening will be randomised in a 1:1 ratio to experimental (combination) arm versus control (mono therapy) arm.

Randomisation will be performed by computer generated random codes (performed by Singapore Clinical Research Institute) with a masked allocation sequence. There will be no blinding of therapy and the study will be conducted as an open label study since the outcomes are objectively measurable.

After randomisation patients will be monitored 12 weekly for the first 24 weeks, then every 24 weekly until the last visit at 96 weeks.

At each visit, patients will have a clinical evaluation and have a panel of laboratory tests:

* Hematology: Full blood count, prothrombin time and international normalized ratio
* Chemistry: Sodium, potassium, creatinine, albumin, alkaline phosphatase, -aspartate transaminase, alanine transaminase, lactate dehydrogenase, total bilirubin, creatine phosphokinase, alphafetoprotein,
* Urinalysis: Urine dipstick (Appearance, color, leucocytes, nitrite, urobilinogen, protein, PH, specific gravity, ketone, bilirubin and glucose).
* Viral serology: HBeAg, anti-HBe, HBsAg, qHBsAg and anti-HBs

ELIGIBILITY:
Inclusion Criteria:

* Presence of positive HBsAg or HBV DNA for at least 6 months.
* Documented HBeAg positive or HBeAg negative.
* On any NA (lamivudine, adefovir, entecavir, tenofovir or combination of any of these four) for ≥ 1 year
* HBV DNA viral load ≤1.0 x 10^5 copies/ml at screening
* ALT ≤ 1 x ULN (upper limit normal) U/L
* A transient elastography (Fibroscan®) to evaluate the fibrosis stage will be performed at screening if it is not done in the past 6 months prior to screening. -Patient with compensated cirrhosis are permitted for this study.
* eGFR ≥ 50 mL/min, as calculated by CKI-EPI equation.
* Patient has agreed not to take any other investigational drug or systemic anti-viral, cytotoxic, corticosteroid, immunomodulatory agents or Chinese traditional remedies unless clinically indicated.
* Patient is able to give written consent prior to study start and to comply with the study requirements.
* Women of childbearing potential age must have a negative serum (ß-HCG) pregnancy test taken within 14 days of starting therapy
* Lactating/breastfeeding female subjects must agree to discontinue nursing before initiation of study medication(s).

Exclusion Criteria:

* Evidence of decompensated liver disease defined as direct (conjugated) bilirubin >1.2xULN, prothrombin time (PT) >1.5x upper limit of normal (ULN), serum albumin <35 g/L, or prior history of clinical hepatic decompensation (egs. ascites, encephalopathy, variceal hemorrhage).
* Evidence of hepatocellular carcinoma (HCC).
* Have any of the following laboratory tests within 4 weeks of study entry:

  * Active co-infection with HIV antibody or HCV antibody or HDV antibody positivity
  * Evidence of chronic renal insufficiency as defined by an eGFR (by CKD-EPI equation of < 50 mL/min).
* Previous treatment with any form of interferon, Immunomodulators, systemic cytotoxic agents, or systemic corticosteroids within 6 months prior to screening.
* Prolonged exposure to known hepatotoxins such as alcohol or drugs.
* History of clinically relevant psychiatric disease, seizures, central nervous system dysfunction, severe pre-existing cardiac, renal, hematological disease or medical illness that in the investigator's opinion might interfere with therapy.
* Current or known history of malignant disease within 5 years of trial entry.
* Patients with a history of or currently known muscle related disease.
* Liver or any other organ transplant other than cornea and hair.
* Women who are pregnant and who are not practicing adequate birth control measures, or who are lactating.
* Patients with specific contraindications to study drugs according to their Singapore Package Insert.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
quantitative HBsAg (qHBsAg) reduction >1 log IU/ml | Baseline to week 96
  Proportion of patients who have a reduction of qHBsAg >1 log IU/ml from baseline to week 96, in experimental arm versus control arm

SECONDARY OUTCOMES:
HBsAg loss | Baseline to week 96
  Proportion of patients who achieve HBsAg loss at week 96 in experimental versus control arms
HBsAg seroconversion | Baseline to week 96
  Proportion of patients who achieve HBsAg seroconversion at week 96 in experimental versus control arms
HBeAg loss | Baseline to week 96
  Proportion of patients who achieve HBeAg loss at week 96 in experimental versus control arms
HBeAg seroconversion | Baseline to week 96
  Proportion of patients who achieve HBeAg seroconversion at week 96 in experimental versus control arms
quantitative HBsAg decline by >0.5 log10 IU/mL | Baseline, week 24, 48 and 96
  Proportion of patients who have a reduction of qHBsAg >0.5 log IU/ml from baseline to week 96, in experimental arm versus control arm
Alteration in eGFR | Baseline to week 96
  Proportion of patients who have an increase in eGFR from baseline to week 96, in experimental arm versus control arm

CONTACTS AND LOCATIONS:
Overall Officials: Seng Gee Lim, MBBS, FRACP, FRCP, MD, FAMS, Principal Investigator — National University Health System
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] European Association For The Study Of The Liver. EASL clinical practice guidelines: Management of chronic hepatitis B virus infection. J Hepatol. 2012 Jul;57(1):167-85. doi: 10.1016/j.jhep.2012.02.010. Epub 2012 Mar 20. No abstract available. PMID 22436845
- [Background] Piratvisuth T, Komolmit P, Tanwandee T, Sukeepaisarnjaroen W, Chan HL, Pessoa MG, Fassio E, Ono SK, Bessone F, Daruich J, Zeuzem S, Cheinquer H, Pathan R, Dong Y, Trylesinski A. 52-week efficacy and safety of telbivudine with conditional tenofovir intensification at week 24 in HBeAg-positive chronic hepatitis B. PLoS One. 2013;8(2):e54279. doi: 10.1371/journal.pone.0054279. Epub 2013 Feb 4. PMID 23390496
- [Background] Liaw YF. Clinical utility of hepatitis B surface antigen quantitation in patients with chronic hepatitis B: a review. Hepatology. 2011 Aug;54(2):E1-9. doi: 10.1002/hep.24473. PMID 21793018
- [Background] Chan HL, Thompson A, Martinot-Peignoux M, Piratvisuth T, Cornberg M, Brunetto MR, Tillmann HL, Kao JH, Jia JD, Wedemeyer H, Locarnini S, Janssen HL, Marcellin P. Hepatitis B surface antigen quantification: why and how to use it in 2011 - a core group report. J Hepatol. 2011 Nov;55(5):1121-31. doi: 10.1016/j.jhep.2011.06.006. Epub 2011 Jun 28. PMID 21718667
- [Background] Wursthorn K, Jung M, Riva A, Goodman ZD, Lopez P, Bao W, Manns MP, Wedemeyer H, Naoumov NV. Kinetics of hepatitis B surface antigen decline during 3 years of telbivudine treatment in hepatitis B e antigen-positive patients. Hepatology. 2010 Nov;52(5):1611-20. doi: 10.1002/hep.23905. PMID 20931556
- [Background] Gane EJ, Deray G, Liaw YF, Lim SG, Lai CL, Rasenack J, Wang Y, Papatheodoridis G, Di Bisceglie A, Buti M, Samuel D, Uddin A, Bosset S, Trylesinski A. Telbivudine improves renal function in patients with chronic hepatitis B. Gastroenterology. 2014 Jan;146(1):138-146.e5. doi: 10.1053/j.gastro.2013.09.031. Epub 2013 Sep 22. PMID 24067879
- [Background] Gara N, Zhao X, Collins MT, Chong WH, Kleiner DE, Jake Liang T, Ghany MG, Hoofnagle JH. Renal tubular dysfunction during long-term adefovir or tenofovir therapy in chronic hepatitis B. Aliment Pharmacol Ther. 2012 Jun;35(11):1317-25. doi: 10.1111/j.1365-2036.2012.05093.x. Epub 2012 Apr 16. PMID 22506503